CLINICAL TRIAL: NCT04227990
Title: Plinabulin vs. Pegfilgrastim in Reducing the Duration of Severe Neutropenia in Breast Cancer Patients Receiving Myelosuppressive Chemotherapy With Docetaxel, Doxorubicin, and Cyclophosphamide (TAC)
Brief Title: Plinabulin iv Solution in Prevention of TAC Induced Neutropenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeyondSpring Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BPI-2358-106 Phase 2
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Chemotherapy-induced Neutropenia
MeSH Terms: interventions — NPI 2358; pegfilgrastim; Docetaxel; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- TAC + Pegfilgrastim (6 mg) (Active Comparator)
  Interventions: Drug: Pegfilgrastim; Drug: Docetaxel, doxorubicin, and cyclophosphamide (TAC)
- TAC + Plinabulin 10 mg/m^2 (Experimental)
  Interventions: Drug: Plinabulin; Drug: Docetaxel, doxorubicin, and cyclophosphamide (TAC)
- TAC + Plinabulin 20 mg/m^2 (Experimental)
  Interventions: Drug: Plinabulin; Drug: Docetaxel, doxorubicin, and cyclophosphamide (TAC)
- TAC + Plinabulin 30 mg/m^2 (Experimental)
  Interventions: Drug: Plinabulin; Drug: Docetaxel, doxorubicin, and cyclophosphamide (TAC)
- TAC + Pegfilgrastim (1.5 mg) + Plinabulin (20 mg/m^2) (Experimental)
  Interventions: Drug: Plinabulin; Drug: Pegfilgrastim; Drug: Docetaxel, doxorubicin, and cyclophosphamide (TAC)
- TAC + Pegfilgrastim (3 mg) + Plinabulin (20 mg/m^2) (Experimental)
  Interventions: Drug: Plinabulin; Drug: Pegfilgrastim; Drug: Docetaxel, doxorubicin, and cyclophosphamide (TAC)
- TAC + Pegfilgrastim (6 mg) + Plinabulin (20 mg/m^2) (Experimental)
  Interventions: Drug: Plinabulin; Drug: Pegfilgrastim; Drug: Docetaxel, doxorubicin, and cyclophosphamide (TAC)

INTERVENTIONS:
Drug: Plinabulin — Plinabulin (BPI-2358) is a synthetic, low molecular weight, new chemical entity that belongs to the diketopiperazine class of compounds. Plinabulin is intended for intravenous (IV) infusion and is diluted in D5W and administered for 30 minutes (± 5 minutes).
  Arms: TAC + Pegfilgrastim (1.5 mg) + Plinabulin (20 mg/m^2); TAC + Pegfilgrastim (3 mg) + Plinabulin (20 mg/m^2); TAC + Pegfilgrastim (6 mg) + Plinabulin (20 mg/m^2); TAC + Plinabulin 10 mg/m^2; TAC + Plinabulin 20 mg/m^2; TAC + Plinabulin 30 mg/m^2
Drug: Pegfilgrastim — Pegfilgrastim is a long-acting granulocyte colony-stimulating factor that stimulates the growth of neutrophils, to reduce the incidence of fever and infection in patients with certain types of cancer who are receiving chemotherapy that affects the bone marrow.
  Other Names: Neulasta
  Arms: TAC + Pegfilgrastim (1.5 mg) + Plinabulin (20 mg/m^2); TAC + Pegfilgrastim (3 mg) + Plinabulin (20 mg/m^2); TAC + Pegfilgrastim (6 mg); TAC + Pegfilgrastim (6 mg) + Plinabulin (20 mg/m^2)
Drug: Docetaxel, doxorubicin, and cyclophosphamide (TAC) — Docetaxel is a type of chemotherapy medicine called an taxane. Doxorubicin is a type of chemotherapy medicine called an anthracycline. Cyclophosphamide is a type of chemotherapy medicine called an alkylating agent.

SUMMARY:
The primary purpose of this study is to compare the duration of severe neutropenia (DSN) in patients treated with: Docetaxel, doxorubicin, and cyclophosphamide (TAC) + pegfilgrastim versus Docetaxel, doxorubicin, and cyclophosphamide (TAC) + monotheray plinabulin or combination plinabulin/pegfilgrastim Severe neutropenia is an absolute neutrophil count (ANC) <0.5 × 10^9/L. Docetaxel, doxorubicin, and cyclophosphamide (TAC) will be used as the chemotherapy in this study.

DETAILED DESCRIPTION:
This is a multi-center randomized study, Phase 2 study. 115 patients were enrolled in Phase 2. Two regimens were evaluated in Phase 2: a plinabulin monotherapy regimen and a combination therapy regimen of plinabulin + pegfilgrastim. The monotherapy regimen includes 4 arms: pegfilgrastim 6.0 mg alone; and 10, 20, or 30 mg/m2 plinabulin.

The combination regimen includes 4 arms: pegfilgrastim 6.0 mg alone; and 20 mg/m2 plinabulin + pegfilgrastim 1.5, 3, or 6.0 mg. The pegfilgrastim 6.0 mg alone arm is the control arm for comparison with the monotherapy and combination therapy arms for the interim evaluation.

The purpose of this study is to compare the duration of severe neutropenia (DSN) in patients with early stage (Stage I and II) and Stage III breast cancer (node positive or node negative with high risk of recurrence) receiving docetaxel, doxorubicin, and cyclophosphamide (TAC) and monotherapy plinabulin or combination therapy plinabulin/pegfilgrastim. Severe neutropenia is an absolute neutrophil count (ANC) <0.5 × 10^9/L.

Docetaxel, doxorubicin, and cyclophosphamide (TAC) were used as the chemotherapy in this study. These agents are among the most active and commonly used chemotherapeutic agents employed for treating patients with breast carcinoma.

In particular, TAC chemotherapy has been used for the adjuvant treatment of HER2 negative early breast cancer patients with node positive disease as well as for node negative breast cancer patients who have a high risk of recurrence.

Plinabulin is a novel small molecule that is being developed for the mitigation of chemotherapy-induced neutropenia. Administered by IV infusion on the same day of (approximately 1 hour after) chemotherapy (TAC), plinabulin was given in a single dose per cycle. Plinabulin is being studied to see if it is a convenient alternative to G-CSF, pegfilgrastim, for the prevention of chemotherapy-induced neutropenia.

64 patients were enrolled for monotherapy evaluation and 51 patients were enrolled for the combination therapy Arm 5, 6 and 7 for efficacy and safety evaluation. The arm designation and planned intervention is as follows:

For monotherapy:

Arm 1: TAC + pegfilgrastim (6.0 mg)

Arm 2: TAC + plinabulin (10 mg/m2).

Arm 3: TAC + plinabulin (20 mg/m2).

Arm 4: TAC + plinabulin (30 mg/m2).

For combination therapy:

Arm 1: TAC + pegfilgrastim (6.0 mg)

Arm 5: TAC + plinabulin (20 mg/m2) + pegfilgrastim (1.5 mg)

Arm 6: TAC + plinabulin (20 mg/m2) + pegfilgrastim (3.0 mg)

Arm 7: TAC + plinabulin (20 mg/m2) + pegfilgrastim (6.0 mg)

Cycles 1 to 4 will consist of TAC (or TC for Cycles 2 to 4) administered IV on Day 1, every 21 days. Patients in Arms 2, 3 and 4 will receive a single dose of plinabulin, 30 minutes after the end of the TAC (or TC for Cycles 2 to 4) infusion on Day 1. The plinabulin dose will be infused over 30 minutes (±5 minutes) in Arms 2 and 3 and over 60 minutes (±5 minutes) in Arm 4 (in order to improve tolerability at the higher 30 mg/m2 dose level).

On Day 2 of each cycle (≥24 hours after completing chemotherapy) patients in Arm 1 and in combination therapy will receive a single dose of pegfilgrastim (1.5, 3.0, or 6.0 mg) (subcutaneous injection).

ELIGIBILITY:
Inclusion Criteria:

1. Women who are at least 18 years of age at the time of signing the informed consent form.
2. In the opinion of their treating oncology investigator, are candidates for at least 4 cycles of chemotherapy with TAC (docetaxel, doxorubicin, and cyclophosphamide).
3. Patients who are candidates for adjuvant or neoadjuvant TAC will meet all of the following criteria:

   Biopsy proven, early stage (Stage I and II) and Stage III breast cancer, and Are within 60 days of a diagnostic or surgical procedure (biopsy, umpectomy, mastectomy), and Have had no prior chemotherapy.
4. Pathological confirmation of cancer is required.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Have life expectancy of 3 months or more.
7. The following laboratory results provided by the central laboratory within 14 days prior to study drug administration:

   ANC ≥ 1.5 x 10^9/L independent of growth factor support; hemoglobin ≥ 9 g/dL independent of transfusion or growth factor support; calculated creatinine clearance (CLcr) ≥ 60 mL/min using Cockcroft-Gault formula; Serum total bilirubin ≤ upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) as 2.5 x ULN (≤ 1.5 x ULN if alkaline phosphate is > 2.5 x ULN).
8. Prothrombin time (PT) and International Normalized Ratio (INR) ≤1.5 × ULN, activated partial thromboplastin time (PTT) ≤1.5 × ULN, based on central laboratory results.
9. Women of childbearing potential have a negative pregnancy test at screening. Women of childbearing potential are defined as sexually mature women without prior hysterectomy or who have had any evidence of menses in the past 12 months. However, women who have been amenorrhoeic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti-estrogens, or ovarian suppression.

Women of childbearing potential (i.e., menstruating women) must have a negative urine pregnancy test (positive urine tests are to be confirmed by serum test) documented within the 24-hour period prior to the first dose of study drug.

Sexually active women of childbearing potential enrolled in the study must agree to use two forms of accepted methods of contraception during the course of the study and for 3 months after their last dose of study drug. Effective birth control includes (a) intrauterine device plus one barrier method; (b) on stable doses of hormonal contraception for at least 3 months (e.g., oral, injectable, implant, transdermal) plus one barrier method; (c) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm); or (d) a vasectomized partner.

Exclusion Criteria:

1. History of myelogenous leukemia, myelodysplastic syndrome, or sickle cell disease.
2. Use of strong CYP3A4, CYP2D6 or P-glycoprotein (P-gp) inhibitors and inducers, within 14 days of the first administration of study drug and for the duration of the study.
3. Received an investigational agent or tumor vaccine within 2 weeks before the first dose of study drug; patients must have recovered from toxicity of prior treatment and have no >Grade 1 Common Terminology Criteria for Adverse Events (CTCAE) (v4.03) treatment emergent adverse events (TEAE).
4. Receiving any concurrent anticancer therapies (including concomitant anti-HER2/neu agents such as trastuzumab [Herceptin], trastuzumab emtansine [TDM-1, Kadcyla®], pertuzumab [Perjeta®], lapatinib [Tykerb®]).
5. Received a prior bone marrow or stem cell transplant.
6. Have a co-existing active infection or received systemic anti-infective treatment within 72 hours before the first dose of study drug.
7. Concurrent or prior radiation therapy within 4 weeks before the first dose of study drug.
8. Chronic use of filgrastim, pegfilgrastim, or any bioequivalent (biosimilar) for severe chronic neutropenia or other chronic neutropenia syndrome.
9. Presence of any serious or uncontrolled illness including, but not limited to: uncontrolled diabetes, ongoing or active infection, symptomatic congestive heart failure unstable angina pectoris, uncontrolled cardiac arrhythmia, uncontrolled arterial thrombosis, symptomatic pulmonary embolism, and psychiatric illness that would limit compliance with study requirements or any other conditions that would preclude the patient from study treatment as per the discretion of the Investigator.
10. Significant prior doxorubicin (>240 mg/m2) or anthracycline exposure that would preclude the safe administration of TAC chemotherapy as described in the protocol.
11. Significant cardiovascular history:

    Cardiac ventricular dysfunction inhibiting the patient"s ability to receive 4 cycles of doxorubicin.

    History of myocardial infarction or ischemic heart disease within 1 year (within a window of up to 18 days less than 1 year) before first study drug administration Uncontrolled arrhythmia History of congenital QT prolongation Electrocardiogram (ECG) findings consistent with active ischemic heart disease New York Heart Association Class III or IV cardiac disease; Uncontrolled hypertension: blood pressure consistently >150 mm Hg systolic and > 100 mm Hg diastolic in spite of antihypertensive medication
12. History of hemorrhagic diarrhea, inflammatory bowel disease, or active uncontrolled peptic ulcer disease. (Concomitant therapy with ranitidine or its equivalent and/or omeprazole or its equivalent is acceptable). History of ileus or other significant gastrointestinal disorder known to predispose to ileus or chronic bowel hypomotility.
13. Any other active malignancy requiring active therapy.
14. Known human immunodeficiency virus (HIV) seropositivity.
15. Active Hepatitis B virus (HBV) infection which requires antiviral treatment or the patient has detectable Hepatitis B surface Antigen (HBsAg); hepatitis B surface antibody (anti-HBs) without detectable HBsAg does not exclude patients from the study. Hepatitis C infection (Hepatitis C antibody reactive) which requires treatment also excludes patients from the study.
16. Female patient who is pregnant or lactating.
17. Use of prophylactic antibiotics.
18. Unwilling or unable to comply with procedures required in this protocol.
19. History of allergy to any of the study drugs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 115 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2019-01-03 (Actual)

PRIMARY OUTCOMES:
Duration of Severe Neutropenia (DSN) | Cycle 1 (21 days)
  Days with Severe Neutropenia in treatment Cycle 1

SECONDARY OUTCOMES:
Frequency of Grade 4 neutropenia | Cycle 1 (21 days)
  Frequency of patients with at least 1 day of Grade 4 neutropenia (ANC <0.5 × 109/L)
Bone pain score | Cycle 1 (21 days)
  Mean pain score from the patient bone pain scale from pre-dose Day 1 to Day 8 in Cycle 1 (0-10 scale, higher score means worse outcome)
Change in bone pain score | Cycle 1 (21 days)
  Change in bone pain score from pre-dose Day 1 through Day 8 in Cycle1 (0-10 scale, higher score means worse outcome)
Adverse events | Cycle 1 - 4 (21-day cycle)
  Incidences, occurrences, and severity of AEs/SAEs Cycle 1-4

CONTACTS AND LOCATIONS:
Locations (11):
- China (5):
  - Cancer Center of Guangzhou Medical University Breast Oncology, Guangzhou, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin, Harbin
  - Fourth Hospital of Hebei Medical University Breast cancer department, Shijiazhuang, Hebei
  - China-Japan Union Hospital of Jilin University Tumor department of Hematology, Changchun, Jilin
  - Liaoning Cancer Hospital & Institute, Shenyang, Shenyang
- Ukraine (6):
  - Dnipropetrovsk City Multifunctional Hospital #4 Oncology Department, Dnipro
  - Prykarpatskiy Regional Oncological Center, Ivano-Frankivsk
  - "V.T. Zaycev Institute of General and Urgent Surgery NAMS of Ukraine Dept. of Oncology, Kharkiv
  - Kirovograd Regional Oncological Center, Kropyvnytskyi
  - Public Institution Kryvyi Rih Oncology Center, Krutyi Bereh
  - Odessa regional clinical hospital Thoracic Surgery Department Academician Zabolotnoho, Odesa